CLINICAL TRIAL: NCT04164407
Title: Keratoconus, Corneal Diseases and Transplant Registry (KCDTR)
Brief Title: Keratoconus, Corneal Diseases and Transplant Registry
Acronym: KCDTR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0500
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Corneal Diseases; Keratoconus; Corneal Ulcer; Corneal Trauma; Corneal Dystrophies
Keywords: Pseudophakic and aphakic bullous keratopathy; Ophthalmology; Cornea; Keratoconus; Cornea transplant; Corneal dystrophies; Crosslinking
MeSH Terms: conditions — Corneal Diseases; Keratoconus; Corneal Ulcer; Corneal Injuries; Corneal Dystrophies, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The cornea is the clear layer in front of the iris and pupil. It protects the iris and lens and helps focus light on the retina. Corneal diseases are serious conditions that can cause clouding, distortion, scarring and eventually blindness. There are several types of corneal disease with keratoconus being one of the most prominent.

Keratoconus is a weakening and thinning of the central cornea. This thinking causes the cornea to develop a cone-shaped deformity leading to vison loss. Keratoconus is usually bilateral affecting people between 10 and 25.

This project aims to collect data on patient suffering with corneal diseases and the treatments they receive, including corneal transplantation, over a period of time during routine clinical practice.

A clinical registry such as this can be a very useful tool to provide a real-world view of clinical practice, patient outcomes, safety, and comparative effectiveness.

•Methods:

Data will be collected from the medical records of patients who have suffered from corneal disease and have undergone treatment in the Ophthalmology department of the CHU Montpellier.

A standardized set of data will be collected for all patients. This will include, demographic and social date such as lifestyle and occupation, current and past pathologies and treatment received. This is data that is already collected as part of routine clinical practice.

This will be an ongoing registry with the aim of collecting the maximum data possible. The more patients that are entered and the longer the follow up for each patient, the more valuable the data will become.

•Discussion:

The aim of this registry to help create a better understanding of variations in treatment and outcomes; to examine factors that influence prognosis; to describe treatment patterns, including appropriateness and effectiveness of treatment and disparities in the delivery of care; to monitor safety and harm and to measure quality of care.

In the long term the data collected in the registry may serve as a basis for the development of evidence-based clinical management guidelines to help clinicians deliver the most appropriate treatment for corneal diseases in the safest and most efficient manner.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from a corneal disease
* Undergoing treatment in the Ophthalmology department of the CHU Montpellier
* Has been presented with an Opt-Out consent form

Exclusion Criteria:

* Expressed a desire to not be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with corneal disease, including keratoconus and / or corneal transplant.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | 1 day
  Visual Acuity

SECONDARY OUTCOMES:
Treatment(s) received | 1 day
  Treatment(s) received

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Daien, MD, PhD, HDR, Study Director — University Hospitals of Montpellier
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC